CLINICAL TRIAL: NCT03230279
Title: Randomized Controlled Trial Of Minimally Invasive Sacroiliac Joint Fusion Compared To Radiofrequency Ablation For Sacroiliac Joint Dysfunction
Brief Title: Sacroiliac Joint Fusion Comparison Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was not financed, Sponsor withdrawn
Sponsor: Ochsner Health System (Other)
Collaborators: Globus Medical Inc (Industry)
Responsible Party: Principal Investigator, Daniel Denis, Neurosurgeon staff at Ochsner Medical Center and Clinical Assistant Professor, Dept. Neurosurgery, Tulane University School of Medicine, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X-99
Record Dates: First submitted 2017-07-18; First posted 2017-07-26 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Sacroiliac Joint Somatic Dysfunction; Sacroiliac; Spondylitis
Keywords: Sacroiliac pain; Low back pain
MeSH Terms: conditions — Spondylitis; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Study Population: Chronic SIJ dysfunction patients presenting at selected Ochsner Health System healthcare centers
  Recruiting mode: Participation will be offered by the principal investigator or the sub-investigators during an outpatient visit in the neurosurgery or pain management clinic.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacroiliac joint fusion (Active Comparator): The subject will receive a sacroiliac joint fusion
  Interventions: Procedure: Sacroiliac joint fusion
- Sacroiliac radio frequency ablation (Active Comparator): The subject will receive a sacroiliac joint radiofrequency ablation
  Interventions: Procedure: Sacroiliac joint radiofrequency ablation

INTERVENTIONS:
Procedure: Sacroiliac joint fusion — Minimally invasive SIJ fusion will be performed under general anesthesia with fluoroscopy. Using SI-LOK®, Sacroiliac Joint Fixation System, Globus Medical Inc. (Audubon, PA), this procedure involve placement of 2 to 3 implants across the SIJ to achieve stabilization and arthrodesis.
  Other Names: Minimally invasive sacroiliac joint arthrodesis
  Arms: Sacroiliac joint fusion
Procedure: Sacroiliac joint radiofrequency ablation — Sacroiliac joint radio frequency ablation will be performed using either conventional or cooled radiofrequency ablation techniques aimed at the S1-S3 lateral branches and the L5 dorsal ramus. The choice between conventional or cooled RFN will be determined by the provider expertise.
  Other Names: Sacroiliac joint neurotomy
  Arms: Sacroiliac radio frequency ablation

SUMMARY:
Patients diagnosed with chronic SIJ pain that can be treated by sacroiliac joint fusion or radiofrequency ablation. The radio frequency ablation is performed using either conventional or "cooled" techniques aimed at the S1-S3 lateral branches and the L5 dorsal ramus. Minimally invasive sacroiliac joint consists of implanting 2 to 3 metallic implants inside the SIJ to increase the stability and eventually fuse the SIJ. This randomized controlled trial aims at comparing treatment success at 6-month follow-up time-point after minimally invasive sacroiliac joint fusion and radiofrequency ablation for chronic SIJ dysfunction.

DETAILED DESCRIPTION:
Introduction This document is a protocol for a human research study. This study is to be conducted according to US and international standards of Good Clinical Practice (FDA Title 21 part 312 and International Conference on Harmonization guidelines), applicable government regulations and Institutional research policies and procedures.

Background

Sacroiliac joint (SIJ) dysfunction is a common pain condition involving the buttock and may irradiate in the low back, groin and/or lower extremity. About one in five patients with low back pain is estimated to have SI joint pain. The economic burden of SIJ pain is high in the United States and there is a need for more cost effective treatment options. There is a lack of relevant high quality studies that compared nonsurgical and surgical treatment for SI joint dysfunction.

Sacroiliac joint (SIJ) dysfunction has been estimated to be the origin of lower back pain in 13 to 30% of patients. SIJ pain is usually referred to the buttock, low back, groin and/or lower extremity. SIJ osteoarthritis, trauma, SIJ degeneration following lumbar fusion and postpartum SIJ dysfunction are common causes of SIJ pain found in a clinical setting. Other less common causes for SIJ pain include inflammatory sacroiliitis, infective sacroiliitis, insufficiency stress fractures and neoplasia.

Diagnostic evidences for SIJ dysfunction

The presenting symptoms of SIJ dysfunction can be similar to those of other spinal conditions such as disc herniation or degenerative spinal stenosis. Unlike radiculopathy, there is often an absence of specific radiological finding with SIJ dysfunction. A gold standard for SI joint pain diagnosis does not exist, but dual comparative local anesthetic joint blocks with at least 70% pain relief are considered a validated diagnostic test for SI joint pain. Reproducibility of SIJ pain with at least 3 SIJ-selective stressing tests, including the thigh trust, compression, Patrick's, distraction and Gaenslen's test, is also considered having good diagnostic validity.

Investigational Agents and Preclinical Data

Nonsurgical treatment efficacy for SIJ dysfunction

Sacroiliac dysfunction is thought to be secondary to a loss of SIJ stability caused by either deficient form closure (joint anatomy) or force closure (compressive forces exerted by neuromuscular and ligamentous structures around the joint. Physical therapy can improve SI joint pain by increasing force closure. Pelvic stabilization, strengthening and self-bracing exercises have been showed to improve force closure and may provide SIJ pain relief.

When SIJ pain fails to improve with physical therapy, several pain management interventions can be offered to patients. Up to now, the level of evidence for SIJ intraarticular or periarticular steroid injections is mainly limited to short-term outcome (3 months) and the effectiveness results are conflicting between different studies.

Compared to conventional radio frequency ablation, the effectiveness of cooled radiofrequency ablation is supported by superior level of evidence. Two randomized controlled trials comparing cooled radio frequency ablation vs placebo demonstrated a success rate varying between 38 to 57% at 6 months for cooled radiofrequency ablation. Observational studies also demonstrated success rate varying from 40% to 71% at 6 months for both conventional and cooled radio frequency ablation. The effectiveness of conventional and cooled radio frequency ablation at 9 and 12 months are more limited and some studies did report loss of effectiveness at 12 months. Based on the available data, there is no evidence supporting clinical superiority between traditional and cool radio frequency ablation. A retrospective study on 88 patients revealed comparable effectiveness between conventional and cool radio frequency ablation with > 50% pain reduction in the majority of patients after 3 and 6 months.

Surgical treatment evidence for SIJ dysfunction

Minimally invasive SIJ fusion is a surgical treatment aimed at stabilizing the SIJ to reduce pain, disability and improve quality of life. In a recent randomized controlled trial called Investigation of Sacroiliac Fusion Treatment (INSITE), minimally invasive SIJ fusion, using triangular titanium implants (iFuse Implant System, SI-BONE®, San Jose, CA), has been shown superior to non-surgical treatments in managing SIJ dysfunction at 6 months (81.4% vs 26.1% success rate) and the results in the surgical group were sustained at one year and two years of follow-up. In this trial, success rate was defined as a decreased in SIJ pain Visual Analogue Score of at least 20 mm compared to baseline, an absence of device-related serious adverse events, an absence of neurological worsening and no surgical reintervention. There were 101 subjects in the SIJ fusion group who completed the 6 months follow-up.

Clinical Data to Date The INSITE study is the first and only published Level 1 randomized controlled trial to have compared SIJ fusion with nonsurgical treatment. Although this study demonstrated prolonged improvement in pain, disability and quality of life with SIJ fusion, superiority of SIJ fusion compared to nonsurgical treatment at 6 months cannot be generalized. This superiority trial may not have been truly clinically relevant because there was no specific treatment protocol used in the nonsurgical group for each subject. Nonsurgical management consisted of physical therapy in 98%, at least one steroid injection in 74%, 2 steroid injections in 4% and radiofrequency ablation of the sacral nerve root lateral branches in 46% of the 46 subjects assigned to nonsurgical treatment. The different proportions of treatment offered in the nonsurgical group may in fact differ from other pain management clinical practices and the generalizability of the results is questionable.

Compared to all nonsurgical treatment available for SIJ pain, the effectiveness of radiofrequency ablation is supported by literature of higher level of evidence. Prolonged therapeutic effect up to 6 months after the procedure has been demonstrated for radiofrequency ablation. In the INSITE study, only 21 subjects received radio frequency ablation, a group size that corresponds to only 21% of the number of subjects studied for SIJ fusion. This may explain why the nonsurgical group only had 26.1% success rate in this trial. The quality of evidence for the INSITE study may also be contested as the study sponsor, SI-BONE®, participated in the manuscript redaction and performed the statistical analysis.

The costs of nonsurgical treatments for SIJ pain are substantial in the United Sates medicare population and there is a need to assess the best cost effective therapy for SI joint pain. SIJ fusion and RFN are two SIJ pain treatment modalities that have been studied with a higher level of evidence compared to other modalities, showing significant effectiveness lasting more than 6 months after each procedure. However the effectiveness and costs associated with these two different treatments have never been compared in a clinically relevant randomized trial.

Dose Rationale and Risk/Benefits

RISKS

General / Unforeseeable

The risks of receiving a SIJ fusion include but are not limited to:

* post-operative incisional pain or worsened pain due to muscle spams
* hematoma and/or surgical site infection (less likely)
* nerve damage that can cause paralysis, loss of sensation or pain (unlikely
* possible second intervention for revision or withdrawal of implants (unlikely)

The risks of receiving SIJ radiofrequency ablation include but are not limited to:

* Pain or discomfort around the area treated
* numbness of skin covering the area treated, worsened pain due to muscle spasm,
* permanent nerve pain (less likely)
* allergies or reactions to medications, infection and/or hematoma (less likely) 3rd degree burn (rare)
* Nerve damage due to trauma (rare)

Other risks that are not specifically related to SIJ fusion or SIJ radiofrequency ablation but may occur during any procedure include:

* cardiovascular and /or cerebrovascular events
* cardiac arrhythmia
* deep vein thrombosis
* pulmonary emboli
* pneumonia
* urinary tract infection
* skin abrasions
* coma or death

Radiation Risks

Fluoroscopy is an imaging technique that uses X-rays during the SIJ fusion or SIJ radiofrequency ablation. This form or ionizing radiation poses a potential for increasing the patient's risk of radiation-induced cancer. Radiations doses and exposure during the study are the same that would be used if the subjects were receiving the treatment outside of this study. Therefore, this study does not involve any additional radiation risk for the subjects.

Study Objectives

Primary objective: Determine clinical superiority between minimally invasive SIJ fusion and radiofrequency ablation in chronic SIJ dysfunction patients

Secondary Objectives: Compare cost-effectiveness between treatment groups

Study Design

General Design

* Randomized controlled trial where randomization is done by a random number generator. Even numbers will be directed to the SI joint procedure group and odd numbers will be directed to the radiofrequency ablation procedure.
* The enrolment uses a 1:1 ratio of SIJ fusion to radio frequency ablation
* The subjects and investigators are not blinded to treatment allocation

Subjects will have a detailed medical history and will complete these questionnaires

* SIJ pain rating using the Visual Analogue Scale (VAS)
* Oswestry Disability Index (ODI)
* Short Form-36 (SF-36)

All subjects will be evaluated at randomization and at follow-up visits scheduled at 1, 3, 6, 9, and 12 months.

ELIGIBILITY:
Once the informed consent has been obtained, the following screening procedures/tests will be performed:

* Local anesthetic sacroiliac joint block and steroid injection performed by a qualified Ochsner pain management provider in less than 3 months following the consent date
* The subject will rate his pain level using the VAS at 2, 4, 6, 8 and 10 hours after the sacroiliac joint block and steroid injection
* Patient will be excluded from the study if they do not meet this criteria: VAS defined as at least 75% pain relief that is sustained for at least 2 hours in a 10 hours period after the block
* Sacroiliac joint injection will be done without any analgesics but anti anxiety medication can be used on case by case based
* The subject will attend a follow-up visit at 6 weeks after the SIJ block and steroid injection. During this visit if the subject's VAS has recurred to at least 50mm the patient will be randomized in either sacroiliac joint fusion or radiofrequency ablation.
* Subjects with VAS smaller than 50mm will be seen at 12 weeks of follow-up. During this visit if the subject's VAS has recurred to at least 50mm the patient will be randomized in either sacroiliac joint fusion or radiofrequency ablation. Subjects with smaller that 50mm VAS will be excluded from randomization at this time point.

Inclusion Criteria:

Participation will be offered by treating physicians during an outpatient visit in the neurosurgery or pain management clinic. Subjects need to meet all inclusion criteria in order to participate in the study.

* Male or female
* Age ≥ 18 years old
* Subject is willing and able to give informed consent for participation in the study
* Unilateral or bilateral SIJ pain for more than 50 days
* Persistent SIJ pain despite a trial of physical therapy for SI joint pain
* Agreement to avoid conception during trial
* Average VAS of at least 50 mm
* Minimal ODI score of at least 40%
* Etiology of SIJ dysfunction: osteoarthritis, past surgical history of lumbar or lumbosacral fusion, traumatic injury, post-partum.
* The SIJ pain can not be explained by a lumbar spine pathology seen on MRI: (disc herniation, lateral recess stenosis, moderate or severe spinal stenosis, synovial cyst, mass)
* Successful SIJ injection based on criteria discussed in recruitment section

Exclusion Criteria:

All participants meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Neurological deficit
* History of cancer
* Active spinal or systemic infection
* Past medical history or active psychiatric condition
* Prohibited drug use
* Subject with pacemaker
* Pregnancy or Breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 6 months after the intervention
  Comparison in the proportion of subjects having a success between groups at 6-month follow-up time-point. Treatment success is defined as a ≥ 50% decrease in VAS pain score; a 10-point increase in SF-36BP (amelioration); a 15-point decrease in ODI (amelioration); absence of device-related serious adverse events; absence of focal neurological deficit or neuropathic pain related to lumbosacral nerve roots injury and absence of surgical reintervention for SIJ pain (revision, removal of hardware, additional fixation)

SECONDARY OUTCOMES:
Cost-effectiveness between SIJ fusion and radio frequency ablation | 6 months after the intervention
  Cost-effectiveness comparison between groups. Cost-effectiveness is measured using the SF-6D utility score
Mean changes from baseline in visual analog score for pain | 6 months after the intervention
  Comparison of mean changes from baseline between groups in VAS
Radiofrequency ablation subgroups analysis | 6 months after the intervention
  Subgroups analysis will be carried on between conventional and cooled radio frequency ablation to attempt to determine if any effect is attributable to one form of RFN or the other
Mean changes from baseline in Oswestry Disability Index score | 6 months after the intervention
  Comparison of mean changes from baseline between groups in ODI score
Mean changes from baseline in SF-36 physical component summary score | 6 months after the intervention
  Comparison of mean changes from baseline between groups in SF-36 physical component summary score
Mean changes from baseline in SF-36 mental component summary score | 6 months after the intervention
  Comparison of mean changes from baseline between groups in SF-36 mental component summary score

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Denis, MD-MSc, Principal Investigator — Ochsner Health System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maigne JY, Aivaliklis A, Pfefer F. Results of sacroiliac joint double block and value of sacroiliac pain provocation tests in 54 patients with low back pain. Spine (Phila Pa 1976). 1996 Aug 15;21(16):1889-92. doi: 10.1097/00007632-199608150-00012. PMID 8875721
- [Background] Schwarzer AC, Aprill CN, Bogduk N. The sacroiliac joint in chronic low back pain. Spine (Phila Pa 1976). 1995 Jan 1;20(1):31-7. doi: 10.1097/00007632-199501000-00007. PMID 7709277
- [Background] Sembrano JN, Polly DW Jr. How often is low back pain not coming from the back? Spine (Phila Pa 1976). 2009 Jan 1;34(1):E27-32. doi: 10.1097/BRS.0b013e31818b8882. PMID 19127145
- [Background] Borowsky CD, Fagen G. Sources of sacroiliac region pain: insights gained from a study comparing standard intra-articular injection with a technique combining intra- and peri-articular injection. Arch Phys Med Rehabil. 2008 Nov;89(11):2048-56. doi: 10.1016/j.apmr.2008.06.006. PMID 18996232
- [Background] Capobianco R, Cher D; SIFI Study Group. Safety and effectiveness of minimally invasive sacroiliac joint fusion in women with persistent post-partum posterior pelvic girdle pain: 12-month outcomes from a prospective, multi-center trial. Springerplus. 2015 Oct 5;4:570. doi: 10.1186/s40064-015-1359-y. eCollection 2015. PMID 26543705
- [Background] Longo UG, Loppini M, Berton A, Laverde L, Maffulli N, Denaro V. Degenerative changes of the sacroiliac joint after spinal fusion: an evidence-based systematic review. Br Med Bull. 2014 Dec;112(1):47-56. doi: 10.1093/bmb/ldu030. Epub 2014 Oct 29. PMID 25355839
- [Background] Unoki E, Abe E, Murai H, Kobayashi T, Abe T. Fusion of Multiple Segments Can Increase the Incidence of Sacroiliac Joint Pain After Lumbar or Lumbosacral Fusion. Spine (Phila Pa 1976). 2016 Jun;41(12):999-1005. doi: 10.1097/BRS.0000000000001409. PMID 26689576
- [Background] Kok HK, Mumtaz A, O'Brien C, Kane D, Torreggiani WC, Delaney H. Imaging the Patient With Sacroiliac Pain. Can Assoc Radiol J. 2016 Feb;67(1):41-51. doi: 10.1016/j.carj.2015.08.001. Epub 2015 Nov 26. PMID 26632100
- [Background] Irwin RW, Watson T, Minick RP, Ambrosius WT. Age, body mass index, and gender differences in sacroiliac joint pathology. Am J Phys Med Rehabil. 2007 Jan;86(1):37-44. doi: 10.1097/phm.0b013e31802b8554. PMID 17304687
- [Background] Simopoulos TT, Manchikanti L, Gupta S, Aydin SM, Kim CH, Solanki D, Nampiaparampil DE, Singh V, Staats PS, Hirsch JA. Systematic Review of the Diagnostic Accuracy and Therapeutic Effectiveness of Sacroiliac Joint Interventions. Pain Physician. 2015 Sep-Oct;18(5):E713-56. PMID 26431129
- [Background] Szadek KM, van der Wurff P, van Tulder MW, Zuurmond WW, Perez RS. Diagnostic validity of criteria for sacroiliac joint pain: a systematic review. J Pain. 2009 Apr;10(4):354-68. doi: 10.1016/j.jpain.2008.09.014. Epub 2008 Dec 19. PMID 19101212
- [Background] Hungerford B, Gilleard W, Hodges P. Evidence of altered lumbopelvic muscle recruitment in the presence of sacroiliac joint pain. Spine (Phila Pa 1976). 2003 Jul 15;28(14):1593-600. PMID 12865851
- [Background] O'Sullivan PB, Beales DJ, Beetham JA, Cripps J, Graf F, Lin IB, Tucker B, Avery A. Altered motor control strategies in subjects with sacroiliac joint pain during the active straight-leg-raise test. Spine (Phila Pa 1976). 2002 Jan 1;27(1):E1-8. doi: 10.1097/00007632-200201010-00015. PMID 11805650
- [Background] Cohen SP, Hurley RW, Buckenmaier CC 3rd, Kurihara C, Morlando B, Dragovich A. Randomized placebo-controlled study evaluating lateral branch radiofrequency denervation for sacroiliac joint pain. Anesthesiology. 2008 Aug;109(2):279-88. doi: 10.1097/ALN.0b013e31817f4c7c. PMID 18648237
- [Background] Patel N, Gross A, Brown L, Gekht G. A randomized, placebo-controlled study to assess the efficacy of lateral branch neurotomy for chronic sacroiliac joint pain. Pain Med. 2012 Mar;13(3):383-98. doi: 10.1111/j.1526-4637.2012.01328.x. Epub 2012 Feb 2. PMID 22299761
- [Background] Cheng J, Pope JE, Dalton JE, Cheng O, Bensitel A. Comparative outcomes of cooled versus traditional radiofrequency ablation of the lateral branches for sacroiliac joint pain. Clin J Pain. 2013 Feb;29(2):132-7. doi: 10.1097/AJP.0b013e3182490a17. PMID 22688606
- [Background] Duhon BS, Cher DJ, Wine KD, Kovalsky DA, Lockstadt H; SIFI Study Group. Triangular Titanium Implants for Minimally Invasive Sacroiliac Joint Fusion: A Prospective Study. Global Spine J. 2016 May;6(3):257-69. doi: 10.1055/s-0035-1562912. Epub 2015 Aug 11. PMID 27099817
- [Background] Polly DW, Cher DJ, Wine KD, Whang PG, Frank CJ, Harvey CF, Lockstadt H, Glaser JA, Limoni RP, Sembrano JN; INSITE Study Group. Randomized Controlled Trial of Minimally Invasive Sacroiliac Joint Fusion Using Triangular Titanium Implants vs Nonsurgical Management for Sacroiliac Joint Dysfunction: 12-Month Outcomes. Neurosurgery. 2015 Nov;77(5):674-90; discussion 690-1. doi: 10.1227/NEU.0000000000000988. PMID 26291338
- [Background] Whang P, Cher D, Polly D, Frank C, Lockstadt H, Glaser J, Limoni R, Sembrano J. Sacroiliac Joint Fusion Using Triangular Titanium Implants vs. Non-Surgical Management: Six-Month Outcomes from a Prospective Randomized Controlled Trial. Int J Spine Surg. 2015 Mar 5;9:6. doi: 10.14444/2006. eCollection 2015. PMID 25785242
- [Background] Ackerman SJ, Polly DW Jr, Knight T, Schneider K, Holt T, Cummings J. Comparison of the costs of nonoperative care to minimally invasive surgery for sacroiliac joint disruption and degenerative sacroiliitis in a United States Medicare population: potential economic implications of a new minimally-invasive technology. Clinicoecon Outcomes Res. 2013 Nov 20;5:575-87. doi: 10.2147/CEOR.S52967. eCollection 2013. PMID 24348055